CLINICAL TRIAL: NCT06367972
Title: A Randomized Phase II Basket Trial EXTENDing Efficacy of Systemic Therapy With Local Consolidative Therapy for OligoProgressive Metastatic Disease (EXTEND-OP)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0070; NCI-2024-03278 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: OligoProgressive Metastatic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NLST Arm (Experimental): Participants are assigned to Group 1, participants will be treated with next-line systemic therapy. The specific next-line systemic therapy will be determined by your doctor.
  - If progression occurs (the disease gets worse), participants may cross over to Group 2 and receive LCT.
  Interventions: Procedure: Next-line Systemic Therapy
- LCT Arm (Experimental): Participants are assigned to Group 2, participants will be treated with LCT and then continue on same systemic therapy participants have been receiving followed by the next line systemic of therapy (if applicable). The specific treatments will be determined by your doctor.
  Interventions: Procedure: Local Consolidation Therapy

INTERVENTIONS:
Procedure: Local Consolidation Therapy — Participants may receive radiation therapy. The choice of LCT and radiation therapy regimen will be determined by a multidisciplinary team including the study doctor.
  Other Names: LCT
  Arms: LCT Arm
Procedure: Next-line Systemic Therapy — The specific next-line systemic therapy will be determined by your doctor.
  Other Names: NLST
  Arms: NLST Arm

SUMMARY:
To find out if local consolidation therapy (such as radiation therapy with or without other local therapies such as surgery, ablation [the removal or destruction of a body part or tissue or its function], or embolization [a procedure that uses particles, such as tiny gelatin sponges or beads, to block a blood vessel]) to all progressive sites of disease can help to control the disease compared with next-line systemic therapy.

DETAILED DESCRIPTION:
Primary Objective:

• To determine whether, in participants with oligoprogressive metastatic disease, LCT to all progressive sites of disease offers a benefit in PFS compared to NLST, across seven tumor types in a basket design.

Secondary Objectives:

* To determine whether LCT improves OS in participants with oligoprogressive disease across seven tumor types.
* To assess safety/tolerability of LCT in participants with oligometastatic disease in tumor subtypes.
* To compare quality of life (QOL) of LCT vs. next-line systemic therapy in participants with oligoprogressive disease.
* To characterize duration and progression-free survival time of participants on same-line systemic therapy (SLST) after LCT in the experimental arm.
* To identify predictive/prognostic biomarkers correlated with a benefit for LCT across tumor types, with the aim being to incorporate these biomarkers into future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Histologically or cytologically confirmed stage IV cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Candidate for LCT (radiation therapy +/- other local therapies such as surgery, ablation, or embolization) to all sites of progressive disease.
* Progressive disease will be defined as a discrete radiologic lesion that has not received prior local therapy. Progressive disease will be defined as RECIST (v1.1) defined progression from pre-baseline imaging to baseline imaging at time of screening for the trial.
* Progressive disease must represent an active lesion, which may be defined as the primary tumor site, regional nodal disease, and/or distant metastatic sites.
* Candidate for radiation therapy to at least one site of disease.
* Between one and five progressive lesions, counted as follows: each lesion (not site) will be counted as one, with the exception of metastatic lymph node stations, which will collectively count as one lesion. Regional nodal stations will be counted as a collective single lesion if oligoprogressive. All progressive lesions must be amenable to local therapy as noted in criterion 4.2.1.5 above.
* Counting of oligoprogressive nodal disease will be based on nodal chains. A nodal chain will be considered a single metastatic lesion if the presence of that node results in the patient as having M1 disease per the TNM staging system, AJCC version 8.0. In addition, one of the following criteria must be met: a) ≥1 LN meets radiologic criteria for metastatic disease via RECIST 1.1 (short axis ≥15mm), b) pathologic assessment has confirmed the presence of metastatic cancer cells, and/or c) the LN exhibits imaging signal characteristic of a metastatic lesion (e.g. FDG avidity, contrast enhancement, etc…). In the event of ambiguity, a study co-Investigator will make a final determination of whether pathologic criteria are met. The following caveats apply:
* In participants with a LN exhibiting a short axis ≥15mm and who have other diagnoses that can produce enlarged LNs (e.g. indolent CLL, sarcoidosis, etc…) or a prior history of benign enlarged LNs will not be considered to have metastatic disease per the discretion of the treating physician.
* LN chains that occur bilaterally will be considered separate metastatic sites. For example, left axilla LNs will counted separately from right axilla LNs.
* The following midline LN chains will be counted as 1 metastatic site: mediastinal, para-aortic, mesenteric.
* The following bilateral LN chains will be counted as 1 metastatic site for unilateral involvement, and 2 for bilateral for involvement: preauricular, cervical and occipital, supraclavicular, infraclavicular, pectoral, axillary, hilar, epitrochlear and brachial, iliac, inguinal and femoral, popliteal.
* Baseline imaging must include a scan done within 4 weeks prior to randomization, demonstrating oligoprogressive disease by RECIST (v1.1) criteria compared to pre-baseline imaging.
* Baseline imaging must be done within 4 weeks prior to randomization, and the following imaging is required: PET/CT scan or CT scan of the chest/abdomen/pelvis. MRI may be substituted as indicated (i.e., CT scan of chest plus MRI abdomen/pelvis). Intracranial imaging is recommended for those histologies/disease sites where intracranial restaging is routinely recommended or appropriate as part of staging/restaging standard-of-care.
* Pre-baseline imaging must be done 6-16 weeks prior to baseline imaging, and it is recommended to have a comparable imaging modality (matched modalities between pre-baseline and baseline imaging). RECIST v1.1 will be utilized to define any progressive sites of disease, and if between 1 and 5 RECIST-defined progressive sites of disease are identified, participant may be eligible. Non-RECIST-eligible lesions may be eligible if radiographic and/or clinical features support this lesion being progressive.
* Participants referred for the study that require immediate LCT can receive treatment to CNS lesions or other symptomatic lesions prior to randomization, but these lesions will be counted towards the total number of oligoprogressive lesions.
* Has one of the following 7 histologic types (metastatic disease): colorectal carcinoma (CRC), renal cell carcinoma (RCC), breast cancer, pancreatic cancer, urothelial (bladder) cancer, prostate cancer, and esophageal cancer.
* Females of childbearing potential must not be breast feeding and must have a negative serum or urine pregnancy test and must agree to use adequate contraception from the time of screening until 3 months after discontinuation of the study medication. Acceptable methods of contraception include total and true sexual abstinence, tubal ligation, hormonal contraceptives that are not prone to drug-drug interactions (IUS Levonorgestrel Intra Uterine System (Mirena), Medroxyprogesterone injections (Depo-Provera)), copper-banded intra-uterine devices, and vasectomized partner. All hormonal methods of contraception should be used in combination with the use of a condom by their sexual male partner. Females of childbearing potential are defined as those who are not surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause). Women will be considered post-menopausal if they have been amenorrheic for the past 12 months without an alternative medical cause. The following age-specific requirements must also apply: Women < 50 years old: they would be considered post-menopausal if they have been amenorrheic for the past 12 months or more following cessation of exogenous hormonal treatments. The levels of Luteinizing Hormone (LH) and Follicle-Stimulating Hormone (FSH) must also be in the post-menopausal range (as per the institution). Women ≥ 50 years old: they would be consider post-menopausal if they have been amenorrheic for the past 12 months or more following cessation of all exogenous hormonal treatments, or have had radiation-induced oophorectomy with the last menses > 1 year ago, or have had chemotherapy-induced menopause with >1 year interval since last menses, or have had surgical sterilization by either bilateral oophorectomy or hysterectomy.
* Non-sterilized males who are sexually active with a female partner of childbearing potential must use adequate contraception for the duration of the study and 3 month after the last dose of study medication. Adequate contraception methods include: birth control pills (eg combined oral contraceptive pill), barrier protection (eg condom plus spermicide, cervical/vault cap or intrauterine device), and abstinence. Participants should not father a child for 6 months after completion of the study medication. Participants should refrain from donating sperm from the start of dosing until 6 months after discontinuing the study medication. If male participants wish to father children they should be advised to arrange for freezing of sperm samples prior to the start of the study medication.
* Demonstration of adequate organ function as defined in the table below, all screening labs to be performed within 4 weeks prior to study enrollment:
* Table of Adequate Organ Function Laboratory Values System Laboratory Value Hematological Absolute neutrophil count (ANC) = ≥500 /mcL Platelets = ≥25,000 / mcL Hemoglobin = ≥7 g/dL Hepatic Serum total bilirubin = ≤ 1.5 mg//dl (except for subjects with Gilbert Syndrome, who may have total bilirubin <3.0 mg/dl) OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 mg/dl AST (SGOT) and ALT (SGPT) = ≤ 3 X ULN OR ≤ 5 X ULN for subjects with liver metastases

Exclusion Criteria:

* Metastatic effusion (e.g. pleural effusion or ascites). Note that participants with an effusion that is too small to sample will be eligible for the trial.
* Leptomeningeal disease.
* Peritoneal carcinomatosis.
* Cognitively impaired subjects (e.g. inability to sign informed consent.)
* Any condition that, in the opinion of the investigator, would interfere with the study treatment or interpretation of the study results.
* Diffuse bone marrow involvement as defined by disease involvement of a BM biopsy from a site that does not have radiologic evidence of a bone metastasis.
* More than 4 prior lines of systemic therapy to treat metastatic disease.
* Diagnosis of active scleroderma, lupus, or other rheumatologic disease which in the opinion of the treating radiation oncologist precludes safe delivery of radiotherapy.
* Known psychiatric or substance abuse disorder/s that would interfere with trial participation.
* Concurrent (synchronous or metachronous) other primary malignancy that in the opinion of the treating physician team presents a substantial risk to the participant's life as a competing risk of death (against the primary oligoprogressive malignancy being considered for LCT as part of this trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2028-10-10 (Estimated); Study Completion 2030-10-10 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Ludmir, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org